CLINICAL TRIAL: NCT06245889
Title: A Pilot Study of Neoadjuvant Response-Adapted Chemotherapy With Pembrolizumab in Patients With Stage 2 and 3 Triple Negative Breast Cancer to Determine Early PET and Biomarker Dynamics
Brief Title: PET Dynamics to Response-Adapted Neoadjuvant Therapy in TNBC
Acronym: NeoADAPT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: J2395; IRB00398141 (Other: JHM IRB)
Record Dates: First submitted 2024-01-23; First posted 2024-02-07 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Triple Negative Breast Cancer
Keywords: breast cancer; triple negative; neoadjuvant
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — Paclitaxel; Carboplatin; pembrolizumab; Doxorubicin; Cyclophosphamide; olaparib; Capecitabine

STUDY DESIGN:
Intervention Model Description: Eligible patients with stage 2 and 3 TNBC (ER<10% eligible) will be treated with 4 cycles of paclitaxel/carboplatin/pembrolizumab prior to surgery. A PET scan will be performed at baseline and after 1 cycle of therapy. A breast MRI will be performed after treatment completion. Patients with complete clinical response will proceed to surgery. Patients with RD will complete neoadjuvant rescue with 4 cycles of doxorubicin/cyclophosphamide prior to surgery. If residual disease identified after surgery, adjuvant therapy to be determined by the treating oncologist (may include doxorubicin/cyclophosphamide/pembrolizumab, capecitabine etc).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant therapy (Experimental): 4 cycles of paclitaxel/carboplatin/pembrolizumab
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Pembrolizumab; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Olaparib; Drug: Capecitabine

INTERVENTIONS:
Drug: Paclitaxel — chemotherapy
  Other Names: Taxol
Drug: Carboplatin — chemotherapy
  Other Names: Paraplatin
Drug: Pembrolizumab — immunotherapy
  Other Names: Keytruda
Drug: Doxorubicin — additional chemotherapy - neoadjuvant or adjuvant rescue
  Other Names: Adriamycin
Drug: Cyclophosphamide — additional chemotherapy - adjuvant rescue
  Other Names: Cytoxan
Drug: Olaparib — adjuvant rescue
  Other Names: Lynparza
Drug: Capecitabine — adjuvant rescue
  Other Names: Xeloda

SUMMARY:
Eligible patients with stage 2 and 3 triple negative breast cancer will be treated with 4 cycles of neoadjuvant paclitaxel/carboplatin/pembrolizumab. A PET scan will be performed at baseline and after 1 cycle of therapy. A breast MRI will be performed after treatment completion. Patients with complete clinical response will proceed to surgery. Patients with clinical residual disease will complete neoadjuvant rescue with 4 cycles of doxorubicin/cyclophosphamide prior to surgery. If residual disease identified after surgery, adjuvant therapy to be determined by the treating oncologist (may include doxorubicin/cyclophosphamide/pembrolizumab, capecitabine etc).

DETAILED DESCRIPTION:
Eligible participants will undergo baseline procedures including research bloodwork, MRI and PET scan. Participants will then be treated with one cycle of paclitaxel, carboplatin and pembrolizumab (TCarbo/pembro). At the end of Cycle one patients will undergo repeat procedures (bloodwork and PET scan), and then continue with treatment for an additional three cycles. ctDNA will be collected on day 1 of each cycle. At the end of treatment patients will undergo repeat MRI.

Patients achieving a clinical complete response (CR) on MRI will proceed with surgery. Patients with clinical residual disease (RD) on MRI will be recommended a biopsy, and be recommended "rescue" neoadjuvant doxorubicin and cyclophosphamide with pembrolizumab (AC/pembro) for four additional cycles, and then proceed with surgery. Note: patients/treating physician may opt to proceed with surgery.

Archival tissue will be collected from the surgical product. Patients achieving a pathologic CR (pCR) may proceed with adjuvant pembrolizumab per standard of care, and treating physician's discretion. Patients with pathological RD may proceed with "rescue" adjuvant AC/pembrolizumab for four additional cycles (if not given neoadjuvantly), per treating physician discretion. The participants may also receive Aadjuvant capecitabine or olaparib as indicated and per treating physician's discretion.

ELIGIBILITY:
Inclusion Criteria:

1. Stage II-III TNBC - estrogen receptor (ER) and progesterone receptor (PR) up to and including 10% is eligible
2. Age ≥ 18 years
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
4. Eligible for standard chemo-immunotherapy as determined by treating physician, including consideration of:

   1. Adequate marrow and organ function
   2. Co-morbid conditions do not preclude the use of chemo-immunotherapy (such as uncontrolled autoimmune disease, or the use of immunosuppressive medications)
5. Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on study

Exclusion Criteria:

1. Patients unable to undergo PET or MRI
2. Evidence of metastatic disease or loco-regional recurrence (i.e. distant or chest wall recurrence)
3. Inflammatory breast cancer
4. Previous treatment with paclitaxel, carboplatin, or immune checkpoint inhibitors

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
SULmax in relation to pCR | 8 months
  Evaluate if lack of decrease in fluorodeooxyglucose (FDG) / positron emission tomography (PET) standardized uptake value corrected for lean body mass (SULmax) by <40% after 1 cycle of neoadjuvant therapy correlates with residual disease at the time of surgery.

SECONDARY OUTCOMES:
Pathologic complete response (pCR) | 3 years
  Evaluate the pathologic complete response (pCR) rate in patients with early-stage triple negative breast cancer (TNBC) treated with neoadjuvant chemo-immunotherapy.
Circulating tumor deoxyribonucleic acid (ctDNA) clearance | 3 years
  Evaluate how circulating tumor deoxyribonucleic acid (ctDNA) kinetics collected at pre-treatment, and during and after completion of neoadjuvant treatment correlate with pathologic complete response (pCR) at the time of surgery.

OTHER OUTCOMES:
Pathologic complete response (pCR) comparison | 3 years
  Compare the pathologic complete response (pCR) rates among patients who achieved clinical complete response (cCR) by breast magnetic resonance imaging (MRI) and those received "rescue" neoadjuvant AC/pembrolizumab with clinical residual disease (RD) after MRI scan.
Diagnostic accuracy of percent and absolute change between baseline and C1D15 measurements | 3 years
  Evaluate the diagnostic accuracy of percent and absolute change (between baseline and C1D15 measurements), and C1D15 absolute measurements in fluorodeooxyglucose (FDG) / positron emission tomography (PET) standardized uptake value corrected for lean body mass (SULmax) for predicting clinical complete response (cCR) using receiver operating characteristic (ROC) curve.
Clinical complete response (cCR) and pathologic complete response (pCR) | 3 years
  Investigate if clinical complete response (cCR) by MRI is predictive of pathologic complete response (pCR).
Change in microbiome | 3 years
  Number of patients that experienced changes in the microbiome serially over time of residual disease.

CONTACTS AND LOCATIONS:
Overall Officials: Cesar A Santa-Maria, MD, Study Chair — Johns Hopkins University
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schmid P, Cortes J, Pusztai L, McArthur H, Kummel S, Bergh J, Denkert C, Park YH, Hui R, Harbeck N, Takahashi M, Foukakis T, Fasching PA, Cardoso F, Untch M, Jia L, Karantza V, Zhao J, Aktan G, Dent R, O'Shaughnessy J; KEYNOTE-522 Investigators. Pembrolizumab for Early Triple-Negative Breast Cancer. N Engl J Med. 2020 Feb 27;382(9):810-821. doi: 10.1056/NEJMoa1910549. PMID 32101663
- [Result] Mittendorf EA, Zhang H, Barrios CH, Saji S, Jung KH, Hegg R, Koehler A, Sohn J, Iwata H, Telli ML, Ferrario C, Punie K, Penault-Llorca F, Patel S, Duc AN, Liste-Hermoso M, Maiya V, Molinero L, Chui SY, Harbeck N. Neoadjuvant atezolizumab in combination with sequential nab-paclitaxel and anthracycline-based chemotherapy versus placebo and chemotherapy in patients with early-stage triple-negative breast cancer (IMpassion031): a randomised, double-blind, phase 3 trial. Lancet. 2020 Oct 10;396(10257):1090-1100. doi: 10.1016/S0140-6736(20)31953-X. Epub 2020 Sep 20. PMID 32966830